CLINICAL TRIAL: NCT04984447
Title: OCT Guided Trans Nasal Imaging of the Small Intestine in Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Guillermo J. Tearney, MD, PhD - Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017P001428
Record Dates: First submitted 2020-08-11; First posted 2021-07-30 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Environmental Enteric Dysfunction
Keywords: EED; Environmental Enteric Dysfunction; Environmental Enteropathy; Tropical Enteropathy; GI; Tethered Capsule Endoscopy; Imaging; Diagnosis
MeSH Terms: conditions — Sprue, Tropical; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Feasibility of TNIB catheter (Experimental): The feasibility of using the TNIB catheter to obtain microscopic images of the intestine. Healthy adult participants, and healthy pregnant women in their 2nd trimester of pregnancy will be enrolled, and their upper gastrointestinal tract will be imaged by the TNIB device
  Interventions: Device: TNIB Catheter

INTERVENTIONS:
Device: TNIB Catheter — Pariticipants will be asked to fast for 8 hours prior to study procedure and no liquids 2 hours prior to study procedure. Lidocaine jelly will may be used to help insert the TNIB Catheter through the Nares. Once inserted past the pharynx, imaging will begin. We will attempt to image the duodenum within 3 hours of study procedure starting.

SUMMARY:
The investigators are seeking healthy adult participants 18-60 years and healthy pregnant women in their 2nd trimester of pregnancy for a research study to assess a new imaging device. The Tearney Laboratory at the Wellman Center for Photomedicine at Massachusetts General Hospital is developing high-resolution imaging devices that can be used to improve diagnostics in gastrointestinal diseases.

DETAILED DESCRIPTION:
The investigators have developed a device that can image the duodenum (the first part of the small intestine). The device consists of a thin, flexible tube with a small internal camera inside of it that takes high-resolution images of the gastrointestinal tract. The device will be introduced through the nose and then advanced into the stomach and duodenum. Participant tolerability, imaging quality and the optimal imaging technique will be evaluated. The results of this study will be used as the basis for a larger study to be conducted at the Aga Khan University Hospital in Pakistan where subjects with suspected or diagnosed EED will be imaged.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Participants who are in their 2nd trimester of pregnancy
* Participant must be 18-60 years of age
* Participant must be able to consent to the procedure.
* Participant must fast (no solid food) for at least 8 hours and have no liquids within 2 hours prior to the procedure.

Exclusion Criteria:

* Participants with a history of upper respiratory disease or surgery
* Pregnant women with high-risk pregnancies such as history of: hyperemesis gravidarum, HIV, severe anemia or any other high-risk pregnancy conditions at the discretion of the subject's physician and the PI
* Participants with a history of upper gastrointestinal surgery
* Pregnant women with Type 1 diabetes
* Pregnant women with Type 2 diabetes on medication and gestational diabetes requiring medication
* Pregnant women with gestational thrombocytopenia
* Participants with upper respiratory infection at least 7 days prior to the procedure
* Pariticipants with any contraindications to the placement of the NJ tube including deviated septum or any other anatomical abnormalities of the nasopharynx or upper gastrointestinal region, history of trans-sphenoidal surgery, facial or cranial trauma and fractures, chronic sinusitis, esophageal strictures, varices etc.
* Participants on medications that delay gastric emptying.
* Participants on drugs which impair clotting like anticoagulants and antiplatelet drugs, NSAIDS, history of bleeding disorders.
* Participants using nasal steroids or any steroids for environmental allergies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Ability for participant to tolerate the device | 3 hours
  Can the participant tolerate the administration of the device with minimal discomfort?
Ability to visualize gastrointestinal features | 6 months
  Can the technology successfully visualize gastrointestinal features?

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States